CLINICAL TRIAL: NCT00567437
Title: Utility of Exercise-induced NT-pro-brain Natriuretic Peptide Levels in Predicting Prognosis in Asymptomatic Aortic Stenosis
Brief Title: Utility of Exercise-induced N-terminal (NT) Pro-brain Natriuretic Peptide Levels in Predicting Prognosis in Asymptomatic Aortic Stenosis
Acronym: AS-BNP
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Poor patient enrollment from clinic secondary to investigator illness.
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Pro00002221
Record Dates: First submitted 2007-12-04; First posted 2007-12-05 (Estimated); Last update posted 2012-10-24 (Estimated); Status verified 2008-11

CONDITIONS: Aortic Stenosis
Keywords: aortic stenosis; prognosis; brain natriuretic peptide
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Other): 10 patients with no aortic stenosis
  Interventions: Other: NT-pro-BNP levels
- B (Other): 100 patients with asymptomatic AS
  Interventions: Other: NT-pro-BNP levels

INTERVENTIONS:
Other: NT-pro-BNP levels — pre- and post-exercise NT-pro-BNP levels

SUMMARY:
One hundred patients with moderate to severe asymptomatic aortic stenosis (AS) will be asked to exercise on a treadmill. NT-pro-BNP levels will be drawn before and after exercise. Changes in NT-pro-BNP levels will be correlated to outcomes at one year. In the pilot phase an additional 10 control subjects without AS will be enrolled to document the control response of NT-pro-BNP elevations with exercise.

ELIGIBILITY:
Inclusion Criteria:

1. valvular AS (Doppler velocity ≥ 3.0 m/s)
2. no baseline symptoms referable to valvular heart disease
3. able to perform ETT

Exclusion Criteria:

1. more than mild aortic regurgitation, mitral regurgitation/ stenosis, or tricuspid regurgitation/stenosis
2. previous AVR
3. known coronary artery disease
4. creatinine clearance 50 mL/min
5. LVEF < 50%
6. planned valve surgery prior to enrollment
7. significant pulmonary disease
8. unable to give informed consent
9. pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2007-12; Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
development of symptomatic aortic stenosis (new/progressive angina or dyspnea, pre-syncope/syncope, hospitalization for cardiac chest pain or heart failure, drop in LV ejection fraction, cardiovascular or sudden death, valve replacement surgery) | one year

CONTACTS AND LOCATIONS:
Overall Officials: Thomas M. Bashore, MD, Principal Investigator — Duke University; John K. Harrison, MD, Principal Investigator — Duke University; Aslan T. Turer, MD, Study Director — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States